CLINICAL TRIAL: NCT02635776
Title: Peanut Allergy Oral Immunotherapy Study of AR101 for Desensitization in Children and Adults (PALISADE)
Acronym: PALISADE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aimmune Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARC003
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Results first posted 2022-03-17 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Peanut Allergy
Keywords: AR101 (Characterized Peanut Allergen); Characterized Peanut Allergen; CPNA (Characterized Peanut Allergen); OIT (oral immunotherapy); Oral Immunotherapy; Peanut Allergy; Allergy; Peanut-Allergic Children; Peanut-Allergic Adults; Desensitization
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity | interventions — Capsules

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AR101 powder provided in capsules & sachets (Experimental): Study product provided as peanut protein in pull-apart capsules or sachets
  Interventions: Biological: AR101 powder provided in capsules & sachets
- Placebo powder provided in capsules & sachets (Placebo Comparator): Placebo formulation in pull-apart capsules or sachets containing only inactive ingredients
  Interventions: Biological: Placebo powder provided in capsules & sachets

INTERVENTIONS:
Biological: AR101 powder provided in capsules & sachets — Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
  Arms: AR101 powder provided in capsules & sachets
Biological: Placebo powder provided in capsules & sachets — Study product formulated to contain only inactive ingredients for use as defined in the protocol
  Arms: Placebo powder provided in capsules & sachets

SUMMARY:
The purpose of this study is to demonstrate the efficacy and safety of AR101 through reduction in clinical reactivity to peanut allergen in peanut-allergic children and adults.

DETAILED DESCRIPTION:
This is an international, multicenter, randomized, double-blind, placebo-controlled study of the efficacy and safety of AR101 in a characterized desensitization oral immunotherapy regimen in peanut-allergic individuals.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 4 through 55 years
* Clinical history of allergy to peanuts or peanut-containing foods
* Serum immunoglobulin E (IgE) to peanut ≥0.35 kUA/L (kilos of allergen-specific units per liter, determined by UniCAP™* within the past 12 months) and/or a skin prick test (SPT) to peanut ≥3 mm compared to control
* Experience dose-limiting symptoms at or before the 100 mg challenge dose of peanut protein (measured as 200 mg of peanut flour) on Screening DBPCFC conducted in accordance with PRACTALL** guidelines
* Not be residing at the same address as another subject in this or any peanut OIT study

UniCAP™*: a laboratory system for routine diagnostic testing of allergy and tool for basic studies on allergens and antibodies

PRACTALL**: PRACTical issues in ALLergology Joint United States/European Union Initiative

Key Exclusion Criteria:

* History of cardiovascular disease, including uncontrolled or inadequately controlled hypertension
* History of severe or life-threatening episode of anaphylaxis or anaphylactic shock within 60 days of Screening DBPCFC
* History of chronic disease (other than asthma, atopic dermatitis, or allergic rhinitis) that is, or is at significant risk of becoming, unstable or requiring a change in chronic therapeutic regimen
* History of eosinophilic esophagitis (EoE), other eosinophilic gastrointestinal disease, chronic, recurrent, or severe gastroesophageal reflux disease (GERD), symptoms of dysphagia or recurrent gastrointestinal symptoms of undiagnosed etiology
* History of severe asthma (NHLBI criteria steps 5 or 6), or mild to moderate asthma (2007 NHLBI criteria steps 1-4) that is uncontrolled or difficult to control
* History of steroid medication use
* History of a mast cell disorder, including mastocytosis, urticarial pigmentosa, and hereditary or idiopathic angioedema
* Developing dose-limiting symptoms in reaction to the placebo part of the Screening DBPCFC
* Having the same place of residence as another subject in the study

Ages: 4 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 555 (Actual)
Dates: Start 2015-12-22 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director of Regulatory Affairs, Study Chair — Aimmune Therapeutics, Inc.
Locations (69):
- United States (49):
  - Banner University of Arizona Medical Center, Tucson, Arizona
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Long Beach Memorial Medical Center / Miller Children's and Women's Hospital, Long Beach, California
  - UCLA Medical Center, Santa Monica, Los Angeles, California
  - Allergy & Asthma Associates of Southern California dba Southern California Research, Mission Viejo, California
  - Sean N. Parker Center for Allergy Research, LPCH at El Camino Hospital, Mountain View, California
  - Peninsula Research Associates, Inc., Rolling Hills Estates, California
  - Allergy & Asthma Medical Group and Research Center, A.P.C, San Diego, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Colorado Allergy & Asthma Centers, P.C., Centennial, Colorado
  - National Jewish Health, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Windom Allergy, Asthma and Sinus, Sarasota, Florida
  - University of South Florida Asthma, Allergy & Immunology Clinical Research Unit, Tampa, Florida
  - Atlanta Allergy & Asthma Clinic, PA, Marietta, Georgia
  - Idaho Allergy LLC dba Idaho Research, Eagle, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Comer Children's Hospital, Chicago, Illinois
  - Sneeze, Wheeze & Itch Associates, LLC, Normal, Illinois
  - IU North Riley Children's Specialists, Carmel, Indiana
  - Chesapeake Clinical Research, Inc., Baltimore, Maryland
  - John Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Clinical Research Institute Inc., Plymouth, Minnesota
  - Children's Mercy on Broadway, Kansas City, Missouri
  - Asthma & Allergy Center, PC, Bellevue, Nebraska
  - Atlantic Research Center, LLC, Ocean City, New Jersey
  - Icahn School of Medicine at Mount Sinai, Clinical Research Unit, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Clinical & Translational Research Center (CTRC), Chapel Hill, North Carolina
  - Clinical Research of Charlotte, Charlotte, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Baker Allergy Asthma & Dermatology Research Center, LLC, Portland, Oregon
  - Children's Hospital of Philadelphia: Allergy / Immunology, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - National Allergy and Asthma Research, LLC, Charleston, South Carolina
  - LeBonheur Children's Hospital - Outpatient Building, Memphis, Tennessee
  - Specially for Children Allergy, Asthma and Immunology Clinic, Austin, Texas
  - Allergy Partners of North Texas Research, Dallas, Texas
  - Children's Medical Center, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Texas Children's Hospital, Houston, Texas
  - Sylvana Research, San Antonio, Texas
  - Virginia Mason Medical Center, Seattle, Washington
  - Northwest Asthma and Allergy Center, Seattle, Washington
- Canada (5):
  - Ohayon, Hamilton, Ontario
  - Cheema Research, Inc., Mississauga, Ontario
  - Ottawa Allergy Research Corp, Ottawa, Ontario
  - Gordon Sussman Clinical Research, Inc., Toronto, Ontario
  - Montreal Children's Hospital, Montreal, Quebec
- Odense Universitetshospital - Department of Dermatology and Allergy Center, Odense, Denmark
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitatsklinikum Frankfurt, Klinik fur Kinger und Jagendmedizin, Frankfurt
  - Medaimun GmbH, Frankfurt am Main
- Cork University Hospital, Cork, Ireland
- Az. Osp. - Univ. degli Studi- Padova, UOSD- Allergie Alimentari,, Padua, Italy
- Netherlands (2):
  - Universitair medisch Centrum Groningen, Groningen
  - University Medical Center Groningen, Groningen
- Spain (3):
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Infantil Universitario Nino Jesus, Madrid
  - Hospital Clinico San Carlos, Madrid
- Barnforskningscentrum, Sachs' Children and Youth Hospital, Stockholm, Sweden
- United Kingdom (3):
  - Guy and St Thomas' NHS Foundation Trust, London
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester
  - University Hospital of South Manchester NHS Foundation Trust, Respiratory and Allergy Clinical Research Facility, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nilsson C, Vereda A, Borres MP, Andersson M, Sodergren E, Rudengren M, Smith A, Simon RJ, Ryan R, Fernandez-Rivas M, Adelman D, Vickery BP. Exploratory immunogenicity outcomes of peanut oral immunotherapy: Findings from the PALISADE trial. Clin Transl Allergy. 2024 Jan;14(1):e12326. doi: 10.1002/clt2.12326. PMID 38282192
- [Derived] Blumchen K, Kleinheinz A, Klimek L, Beyer K, Anagnostou A, Vogelberg C, Butovas S, Ryan R, Norval D, Zeitler S, Du Toit G. Post hoc analysis examining symptom severity reduction and symptom absence during food challenges in individuals who underwent oral immunotherapy for peanut allergy: results from three trials. Allergy Asthma Clin Immunol. 2023 Mar 13;19(1):21. doi: 10.1186/s13223-023-00757-8. PMID 36915184
- [Derived] Nilsson C, Scurlock AM, Dellon ES, Brostoff JM, Pham T, Ryan R, Brown KR, Adelman DC, Aceves SS. Onset of eosinophilic esophagitis during a clinical trial program of oral immunotherapy for peanut allergy. J Allergy Clin Immunol Pract. 2021 Dec;9(12):4496-4501. doi: 10.1016/j.jaip.2021.07.048. Epub 2021 Aug 11. No abstract available. PMID 34389504
- [Derived] Fernandez-Rivas M, Vereda A, Vickery BP, Sharma V, Nilsson C, Muraro A, Hourihane JO, DunnGalvin A, du Toit G, Blumchen K, Beyer K, Smith A, Ryan R, Adelman DC, Jones SM. Open-label follow-on study evaluating the efficacy, safety, and quality of life with extended daily oral immunotherapy in children with peanut allergy. Allergy. 2022 Mar;77(3):991-1003. doi: 10.1111/all.15027. Epub 2021 Sep 24. PMID 34320250
- [Derived] PALISADE Group of Clinical Investigators; Vickery BP, Vereda A, Casale TB, Beyer K, du Toit G, Hourihane JO, Jones SM, Shreffler WG, Marcantonio A, Zawadzki R, Sher L, Carr WW, Fineman S, Greos L, Rachid R, Ibanez MD, Tilles S, Assa'ad AH, Nilsson C, Rupp N, Welch MJ, Sussman G, Chinthrajah S, Blumchen K, Sher E, Spergel JM, Leickly FE, Zielen S, Wang J, Sanders GM, Wood RA, Cheema A, Bindslev-Jensen C, Leonard S, Kachru R, Johnston DT, Hampel FC Jr, Kim EH, Anagnostou A, Pongracic JA, Ben-Shoshan M, Sharma HP, Stillerman A, Windom HH, Yang WH, Muraro A, Zubeldia JM, Sharma V, Dorsey MJ, Chong HJ, Ohayon J, Bird JA, Carr TF, Siri D, Fernandez-Rivas M, Jeong DK, Fleischer DM, Lieberman JA, Dubois AEJ, Tsoumani M, Ciaccio CE, Portnoy JM, Mansfield LE, Fritz SB, Lanser BJ, Matz J, Oude Elberink HNG, Varshney P, Dilly SG, Adelman DC, Burks AW. AR101 Oral Immunotherapy for Peanut Allergy. N Engl J Med. 2018 Nov 22;379(21):1991-2001. doi: 10.1056/NEJMoa1812856. Epub 2018 Nov 18. PMID 30449234

RESULTS

PARTICIPANT FLOW:
Groups:
- AR101: AR101 drug product was supplied in 2 presentations. These were pull-apart capsules containing 0.5, 1, 10, 20 and 100mg of peanut protein and sealed, foil-laminated sachets containing 300mg of peanut protein.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
- Placebo: A Placebo matching the AR101 drug product was supplied in 2 presentations. These were pull-apart capsules matching the 0.5, 1, 10, 20 and 100mg peanut capsules but containing no peanut protein and sealed, foil-laminated sachets matching the peanut protein sachets but without any peanut protein.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
Period: Overall Study
Arm/Group | AR101 | Placebo
Started | 416 | 139
Completed | 314 | 128
Not Completed | 102 | 11
Not completed — Physician Decision | 1 | 0
Not completed — Adverse Event | 51 | 3
Not completed — Withdrawal by Subject | 41 | 7
Not completed — Lost to Follow-up | 4 | 0
Not completed — Other reasons | 5 | 1

BASELINE CHARACTERISTICS:
Population: Measure Analysis Population Description: A total of 555 subjects were enrolled. However, only 551 subjects were included in the intent-to-treat (ITT) population. The ITT Population includes all subjects who received at least one dose of randomized study treatment.
Groups:
- AR101: AR101 drug product provided in two presentations. These were peanut protein in pull-apart capsules or sachets.
  Pull-apart capsules contained 0.5, 1, 10, 20 and 100mg of peanut protein and sealed, foil-laminated sachets contained 300mg of peanut protein.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
- Placebo: A Placebo matching the AR101 drug product was supplied in two presentations. These were pull-apart capsules matching the 0.5, 1, 10, 20 and 100mg peanut capsules but containing no peanut protein and sealed, foil-laminated sachets matching the peanut protein sachets but without any peanut protein.
  The capsules were used during the Initial Escalation and Up-dosing phases of the study. The sachets were used during the Maintenance phase.
- Total: Total of all reporting groups
Arm/Group | AR101 | Placebo | Total
Number analyzed (Participants) | 413 | 138 | 551
Age, Customized [Count of Participants; unit: Participants]
  Age customized categorical: Children (4-11 years) | 238 | 89 | 327
  Age customized categorical: Adolescents (12-17 years) | 134 | 35 | 169
  Age customized categorical: Adults (18-55 years) | 41 | 14 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 180 | 56 | 236
  Male | 233 | 82 | 315
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 17 | 47
  Not Hispanic or Latino | 383 | 121 | 504
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 44 | 10 | 54
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 6 | 3 | 9
  White | 329 | 109 | 438
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 32 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 600 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: The percentage of subjects in the ITT population who achieve desensitization as determined by tolerating specified challenge doses of peanut protein with no more than mild symptoms at the Exit Oral Food Challenge.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Groups:
- AR101: Study product provided as peanut protein in pull-apart capsules or sachets.
  AR101 powder provided in capsules & sachets: Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol
- Placebo: Placebo formulation in pull-apart capsules or sachets containing only inactive ingredients
  Placebo powder provided in capsules & sachets: Study product formulated to contain only inactive ingredients for use as defined in the protocol
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 372 | 124
Participants | 250 | 5
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 600 mg; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 63.2, 95% CI 2-sided [53 to 73.3]

2. Secondary Outcome: Percentage of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 1000 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 372 | 124
Participants | 187 | 3
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 1000 mg; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 47.8, 95% CI 2-sided [38 to 57.7]

3. Secondary Outcome: Percentage of Subjects Ages 4-17 Who Tolerated a Single Highest Dose of at Least 300 mg in the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: as for outcome 1
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 372 | 124
Participants | 285 | 10
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference at 300 mg; Test type: Superiority; p < 0.0001, Farrington-Manning test; Risk Difference (RD) = 68.5, 95% CI 2-sided [58.6 to 78.5]

4. Secondary Outcome: Percentage of Subjects Ages 4-17 by Maximum Severity of Symptoms Occurring at Any Challenge Dose of Peanut Protein During the Exit Double-Blind, Placebo-Controlled Food Challenge (DBPCFC)
Description: The maximum severity of symptoms on 4 levels: 0-None, 1-Mild, 2-Moderate, 3-Severe or higher (Severe, life threatening, fatal) observed in the DBPCFC at any dose (1000 mg or lower).
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | AR101 | Placebo
Number analyzed (Participants) | 372 | 124
Participants
  None | 140 | 3
  Mild | 119 | 35
  Moderate | 94 | 73
  Severe or worse | 19 | 13
Statistical Analysis 1: Comparison: AR101 vs Placebo; Treatment difference in maximum severity; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test (using equally spaced scores), stratified by region (North America, Europe)

ADVERSE EVENTS:
Time Frame: 12 months
Description: The data is presented separately for the 4-17 year old age group (children and adolescents) and 18-55 year old age group (adults).
Groups:
- AR101 (Age 4-17); AR101 (Age 18-55): Study product provided as peanut protein in pull-apart capsules or sachets.
  AR101 powder provided in capsules & sachets: Study product formulated to contain peanut protein at different dosage strengths for use as defined in the protocol.
- Placebo (Age 4-17); Placebo (Age 18-55): Placebo formulation in pull-apart capsules or sachets containing only inactive ingredients.
  Placebo powder provided in capsules & sachets: Study product formulated to contain only inactive ingredients for use as defined in the protocol.
Arm/Group | AR101 (Age 4-17) | Placebo (Age 4-17) | AR101 (Age 18-55) | Placebo (Age 18-55)
All-Cause Mortality (participants affected / at risk) | 0/372 | 0/124 | 0/41 | 0/14
Serious Adverse Events (participants affected / at risk) | 8/372 | 1/124 | 2/41 | 1/14
Other Adverse Events (participants affected / at risk) | 367/372 | 118/124 | 40/41 | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 (Age 4-17) (N=372) | Placebo (Age 4-17) (N=124) | AR101 (Age 18-55) (N=41) | Placebo (Age 18-55) (N=14)
Anaphylactic reaction (Immune system disorders) | 3 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Humerous fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AR101 (Age 4-17) (N=372) | Placebo (Age 4-17) (N=124) | AR101 (Age 18-55) (N=41) | Placebo (Age 18-55) (N=14)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Ear pruritus (Ear and labyrinth disorders) | 25 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 0 | 1 | 1
Eye pruritus (Eye disorders) | 32 | 16 | 0 | 0
Ocular hyperaemia (Eye disorders) | 34 | 10 | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 60 | 17 | 12 | 0
Abdominal pain (Gastrointestinal disorders) | 194 | 30 | 18 | 6
Abdominal pain upper (Gastrointestinal disorders) | 152 | 26 | 16 | 4
Diarrhoea (Gastrointestinal disorders) | 61 | 24 | 13 | 7
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 6 | 1
Dysphagia (Gastrointestinal disorders) | 20 | 3 | 4 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 5 | 1
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Lip pruritus (Gastrointestinal disorders) | 36 | 7 | 4 | 0
Lip swelling (Gastrointestinal disorders) | 38 | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 146 | 29 | 20 | 3
Oral pruritus (Gastrointestinal disorders) | 151 | 20 | 15 | 4
Paraesthesia oral (Gastrointestinal disorders) | 65 | 8 | 15 | 1
Tongue pruritus (Gastrointestinal disorders) | 38 | 7 | 5 | 0
Vomiting (Gastrointestinal disorders) | 154 | 30 | 5 | 3
Asthenia (General disorders) | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 24 | 1 | 3 | 0
Fatigue (General disorders) | 0 | 0 | 3 | 0
Pyrexia (General disorders) | 88 | 27 | 1 | 3
Anaphylactic reaction (Immune system disorders) | 51 | 4 | 7 | 1
Seasonal allergy (Immune system disorders) | 6 | 7 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 24 | 5 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 24 | 7 | 4 | 1
Gastrointestinal viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Impetigo (Infections and infestations) | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 20 | 8 | 3 | 0
Nasopharyngitis (Infections and infestations) | 57 | 20 | 6 | 6
Otitis media (Infections and infestations) | 20 | 5 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 28 | 5 | 1 | 1
Rhinitis (Infections and infestations) | 20 | 11 | 2 | 3
Sinusitis (Infections and infestations) | 16 | 7 | 4 | 2
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 110 | 39 | 9 | 1
Viral infection (Infections and infestations) | 50 | 13 | 3 | 1
Viral upper respiratory tract infection (Infections and infestations) | 15 | 7 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 72 | 28 | 4 | 2
Migraine (Nervous system disorders) | 0 | 0 | 2 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 1 | 1
Renal pain (Renal and urinary disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 42 | 10 | 3 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 152 | 42 | 12 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25 | 2 | 6 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 | 5 | 10 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 80 | 28 | 10 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 70 | 19 | 2 | 3
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Pharyngeal paraesthesia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 6 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 32 | 11 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 113 | 28 | 11 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 98 | 18 | 14 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 152 | 34 | 12 | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 86 | 8 | 12 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 58 | 15 | 7 | 1
Eczema (Skin and subcutaneous tissue disorders) | 32 | 12 | 2 | 1
Erythema (Skin and subcutaneous tissue disorders) | 27 | 5 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 153 | 34 | 16 | 2
Rash (Skin and subcutaneous tissue disorders) | 81 | 18 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 39 | 7 | 3 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 143 | 30 | 12 | 3
Flushing (Vascular disorders) | 49 | 11 | 8 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
* Institutions cannot publish until the multi-center sponsor publication is published
* Or, institutions cannot publish until 18 months after study completion
* And Sponsor review of any publications is required prior to any institution publications according to contractual agreements

DOCUMENTS (2):
  • Study Protocol (2017-07-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT02635776/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT02635776/SAP_001.pdf